CLINICAL TRIAL: NCT04783727
Title: Personalized Therapy Durations Defined by the Blood RNA-based Model for Individualizing Treatment in Multidrug-Resistant Tuberculosis
Brief Title: PredictEndTB Signature for Individualizing Treatment in Multidrug-Resistant Tuberculosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in WHO recommendations for standard of care (control arm); availability of new shorter treatment regimens for MDR-TB; war in Ukraine where two study sites are located; key trial team members left the team.
Sponsor: Research Center Borstel (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PredictEndTBSignature
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Tuberculosis, Pulmonary; Tuberculosis, Multidrug-Resistant; Bacterial Infections; Mycobacterial Infection
Keywords: tuberculosis; multidrug resistance; treatment duration
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis, Multidrug-Resistant; Bacterial Infections; Mycobacterium Infections; Tuberculosis

STUDY DESIGN:
Masking Description: During the treatment, both Participant and Care Provider will be masked but once the treatment end is achieved, they will be unmasked, and study participation is continued.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): The individualised treatment durations defined by the RNA transcriptomic signature-based model
  Interventions: Diagnostic Test: Individualised treatment duration based on RNA transcriptomic model
- Control arm (No Intervention): The locally accepted standard duration of treatment based on the WHO recommendation for treatment of MDR-TB patients

INTERVENTIONS:
Diagnostic Test: Individualised treatment duration based on RNA transcriptomic model — Anti-MDR-TB treatment with standard drugs and individual treatment duration guided by the RNA transcriptomic model; may be shorter or longer than standard WHO-recommended treatment duration of 20 months.
  Arms: Experimental arm

SUMMARY:
PredictEndTB signature is a non-inferiority, prospective, parallel-group open-label randomized controlled trial evaluating the efficacy of individualised antituberculous treatment durations that utilize the transcriptomic signature-based model compared to the standardised twenty months treatment in a cohort of multidrug-resistant tuberculosis patients.

DETAILED DESCRIPTION:
This study is a non-inferiority, prospective, parallel-group open-label randomized controlled trial. Three hundred forty-two HIV-negative patients diagnosed with pulmonary tuberculosis (TB) and starting a new anti-multidrug-resistant tuberculosis (MDR-TB) treatment cycle will be included in the study. Two randomized arms of 171 patients each will be recruited over the two-year period, each patient will be followed-up over the entire course of anti-TB treatment and one year after the end of therapy. Regular study visits will include physical examination, collection of sputum, blood and urine and filling in the study questionnaire. On the collected specimens standard bacteriological and blood tests, as well as extended immunological analysis, will be performed. In the experimental group, an RNA transcriptomic analysis using RNA-Seq technology will also be performed.

In the control arm, the patients will receive a standardised World Health Organization recommended 20 months treatment while in the experimental arm the treatment duration will be guided by the transcriptomic signature-based model.

Treatment outcomes and level of TB relapse and survival within the follow-up period will be compared between the experimental and control arms. The efficacy of biomarker-guided treatment therapy will be assessed by a comparison of the proportions of favourable study outcome between two arms.

ELIGIBILITY:
Inclusion Criteria:

* Patient starting an MDR-TB treatment or within the first 4 weeks after treatment initiation and before culture conversion.
* Rifampicin resistant M. tuberculosis detected in sputum using a nucleic acid amplification test.
* New case of TB or re-treatment.
* Can give informed consent at the point of recruitment.
* Contactable (residing in the area covered by participating TB centres and possessing a landline or a mobile phone).
* Willing to participate for the entire course of the treatment and extensive follow-up.

Exclusion Criteria:

* Age <18 years old.
* Anti-MDR-TB therapy within 6 months prior to the start date of the current treatment cycle.
* HIV infection.
* Non-adherent patient with frequent interruptions.
* Patient in custodianship or guardianship.
* Late exclusion criterion: no positive cultures at inclusion and within the first 3 months of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with favourable study outcome 12 months after treatment end | up to 36 months
  The non-inferiority of the experimental arm compared to the control arm will be established if in the Per-Protocol population the difference in proportions of patients with a favourable study outcome between study arms is greater than the lower equivalence margin of 12%. This outcome measure is assessed after up to 24 months of treatment (usually 20 months) plus 12 months of follow-up after the end of treatment.

SECONDARY OUTCOMES:
Proportion of patients who was lost to follow-up during treatment | up to 24 months
  This outcome measure will be used in the secondary efficacy analysis in the Intention-to-Treat population
Proportion of patients who had a treatment failure | up to 24 months
  This outcome measure will be used in the secondary efficacy analysis in the Intention-to-Treat population
Proportion of patients who died from TB | up to 36 months
  This outcome measure will be used in the secondary efficacy analysis in the Intention-to-Treat population
Proportion of patients who died of any cause | up to 36 months
  This outcome measure will be used in the secondary efficacy analysis in the Intention-to-Treat population

OTHER OUTCOMES:
Proportion of patients experiencing adverse events | up to 24 months
  This outcome measure will be used in the exploratory safety analysis in the safety population
Proportion of patients who experienced TB relapse that was identified on early stages | up to 36 months
  This outcome measure will be used in the safety analysis in the safety population
Characteristics of the transcriptomic signatures obtained at the end of therapy time point and at follow-up visits | up to 36 months
  This outcome measure will be used in the exploratory safety analysis in the safety population

CONTACTS AND LOCATIONS:
Overall Officials: Jan Heyckendorf, MD, Principal Investigator — Research Center Borstel
Locations (5):
- Research Center Borstel, Borstel, Schleswig-Holstein, Germany
- Phthisiopneumology Institute Chiril Draganiuc, Chisinau, Moldova
- Marius Nasta Pulmonology Institute, Bucharest, Romania
- Ukraine (2):
  - Kharkiv National Medical University, Kharkiv
  - National Pirogov Memorial Medical University, Vinnytsia

IPD SHARING:
Plan to Share IPD: No
All study data will be pseudonymised and shared with other researchers only in pseudonymised form

REFERENCES:
- [Background] Heyckendorf J, Marwitz S, Reimann M, Avsar K, DiNardo AR, Gunther G, Hoelscher M, Ibraim E, Kalsdorf B, Kaufmann SHE, Kontsevaya I, van Leth F, Mandalakas AM, Maurer FP, Muller M, Nitschkowski D, Olaru ID, Popa C, Rachow A, Rolling T, Rybniker J, Salzer HJF, Sanchez-Carballo P, Schuhmann M, Schaub D, Spinu V, Suarez I, Terhalle E, Unnewehr M, Weiner J 3rd, Goldmann T, Lange C. Prediction of anti-tuberculosis treatment duration based on a 22-gene transcriptomic model. Eur Respir J. 2021 Sep 2;58(3):2003492. doi: 10.1183/13993003.03492-2020. Print 2021 Sep. PMID 33574078
- [Background] Heyckendorf J, Reimann M, Marwitz S, Lange C; DZIF-TB cohort study group. Pathogen-free diagnosis of tuberculosis. Lancet Infect Dis. 2021 Aug;21(8):1066. doi: 10.1016/S1473-3099(21)00337-6. No abstract available. PMID 34331877